CLINICAL TRIAL: NCT06233955
Title: Effect of Maitland Mobilization With Low Level Laser Therapy in Treatment of Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Kamal Abdel-Shakour, Physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maitland Mobilization and LLLT
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group A received LLLT and Maitland mobilization technique along with conventional physical therapy,
  Interventions: Device: Low Level laser therapy; Other: Maitland mobilization technique
- Group B (Experimental): received LLLT and conventional physical therapy
  Interventions: Device: Low Level laser therapy
- Group C (Experimental): received Maitland mobilization and conventional physical therapy.
  Interventions: Other: Maitland mobilization technique

INTERVENTIONS:
Device: Low Level laser therapy — is a non-invasive light source treatment that generates a single wavelength of light. It emits no heat, sound, or vibration. It is also called photobiology or bio-stimulation
  Other Names: LLLT
  Arms: Group A; Group B
Other: Maitland mobilization technique — is a process of examination; assessment and treatment of musculoskeletal disorders by manipulative physiotherapy where a chain of oscillatory joint mobilization grades based on the pathological limit of tissue are used
  Arms: Group A; Group C

SUMMARY:
Background: Osteoarthritis is a common cause of chronic pain and disability in elderly people.

Objective: To evaluate the efficacy of low-level laser therapy (LLLT) in combination with Maitland mobilization and conventional physical therapy in patients with chronic knee osteoarthritis.

Design: Pre-test post-test randomized control trial.

DETAILED DESCRIPTION:
Knee OA is associated with pain and disability, high treatment costs, decreased productivity, and absence from work and thus has a substantial and growing burden on society Objective: To evaluate the efficacy of low-level laser therapy (LLLT) in combination with Maitland mobilization and conventional physical therapy in patients with chronic knee osteoarthritis.

Participants: Seventy five subjects of both genders with age range from 50 to 65 years, with proven bilateral knee OA diagnosed and referred by orthopaedist were recruited for the study and randomly assigned into three groups.

ELIGIBILITY:
Inclusion Criteria:

Subjects with proven bilateral Knee OA with age range 50- 65 years according to the American College of Rheumatology criteria.

2- Only patients with X-ray stages II and III osteoarthritis selected according to Kellgren & Lawrence classification system.

3- BMI equal to or less than 30 . 4- Patients with Knee pain lasted at least 6 months with intensity at least 3 on VAS scale in activities such as going up-and downstairs, sitting and squatting.

5- Patients with normal mental state. 6- Patients who are not participating in physical therapy in the recent 3 months.

.

Exclusion Criteria:

1. Patient with history of gout, infection, tumour, autoimmune diseases, trauma or other causes of knee pain or knee deformities.
2. Patient with neurologic dysfunction, or with history of chronic disease that may affect the study.
3. Patient with history of knee intra-articular injection in the past 6 months.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | Four weeks
  Is a bidirectional 10 cm straight line with two labels, that is, "no pain" and "worst possible pain", located at either end of the line. Patients were instructed to draw a vertical mark on the line indicating their pain level where zero mean no pain and 10 means worst imaginable pain
Pressure Algometer | Four weeks
  is a handheld pressure algometer that responds linearly to force application between 0 and 5 Kg and it has a 1-cm2 round rubber tip.
Knee digital goniometry | Four weeks
  Baseline digital absolute + axis TM goniometer was used which consisted of one movable arm and one fixed arm and fulcrum

SECONDARY OUTCOMES:
Knee injury and osteoarthritis outcome score short form | Four weeks
  consists of a seven items measure of physical function descended from the items of the function, daily living and function, sports and recreational activity subscales of the KOOS Item responses are coded from 0 to 4, none to extreme respectively. The questionnaire is scored by summing the raw response (range 0-28) and then using the nomogram so the raw score is converted to a true interval score (0-100) where zero means no difficulty and 100 means extreme difficulty

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Cairo university, Cairo, Dokki, Egypt